CLINICAL TRIAL: NCT05803928
Title: Ablation in Combination With Lenvatinib and Anti-PD-1 Antibodies in Patients With Early Recurrence After Radical Resection/Ablation of HCC: a Prospective, Randomized, Controlled Clinical Study
Brief Title: Ablation in Combination With Lenvatinib and Anti-PD-1 Antibodies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hua Li (Other)
Responsible Party: Sponsor-Investigator, Hua Li, Clinical Professor, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2023]02-116-16
Record Dates: First submitted 2023-03-22; First posted 2023-04-07 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ablation + Lenvatinib +anti-PD-1 Antibodies (Experimental): Experimental: ablation + lenvatinib +anti-PD-1 antibodies ablation: ultrasound-guided percutaneous ablation for recurrent hepatocellular carcinoma. After local anesthesia and intravenous sedation, the unipolar needle was gradually inserted into the lesion and placed at the deepest edge of the lesion. Ablation electrodes are unipolar needles with bare ends of 2 or 3cm (depending on tumor size).
  Lenvatinib: (TBILI<2 times the upper limit of normal) about 3 to 7 days after treatment. The dosage and usage of the regimen were 8mg qd po (body weight < 60kg) or 12mg qd po (body weight ≥60kg).
  Anti-PD-1 Antibodies: About 3 to 7 days after radiofrequency ablation, (TBILI<2 times the upper limit of normal). The dosage was used accordingt to the drug instructions., every 3 weeks for a course of treatment. The longest course of treatment is 6 months.
  Interventions: Drug: lenvatinib + anti-PD-1 antibodies; Procedure: ablation
- Ablation (Active Comparator): Experimental group: ablation Ablation: ultrasound-guided percutaneous ablation for recurrent hepatocellular carcinoma. After local anesthesia and intravenous sedation, the unipolar needle was gradually inserted into the lesion and placed at the deepest edge of the lesion. Ablation electrodes are unipolar needles with bare ends of 2 or 3cm (depending on tumor size). The ablation power is 150W (range from 100 to 200W). In general, the average ablation time per lesion is about 12 minutes (ranging from 10 to 15 minutes).
  Interventions: Procedure: ablation

INTERVENTIONS:
Drug: lenvatinib + anti-PD-1 antibodies — A ablation treatment group B ablation+ lenvatinib + anti-PD-1 antibodies treatment group
  Arms: Ablation + Lenvatinib +anti-PD-1 Antibodies
Procedure: ablation — radiofrequency ablation or microwave ablation

SUMMARY:
Lenvatinib is an oral multi-target receptor tyrosine kinase inhibitor (TKI) inhibitor that mainly inhibits the Endothelial growth factor receptor (VEGFR) VEGFR-1,2,3; Fibroblast growth factor receptor, FGFR) FGFR-1,2,3,4; Platelet-derived growth factor receptor (PDGFR) PDGFRα; The kinases RET and KIT, thereby inhibiting tumor cell proliferation, inducing apoptosis, and playing an anti-angiogenic role, have been approved by the FDA and CFDA as first-line treatment for patients with advanced liver cancer. lenvatinib showed longer disease progression than sorafenib (8.9 months vs. sorafenib. 3.7 months), longer progression-free survival (7.4 months vs. 3.7 months), and higher disease control rates (24.1% vs. 9.2%). Therefore, lenvatinib has obvious advantages in HCC treatment because of its strong anti-angiogenic and anti-tumor growth effects.

Cindilimab is a human immunoglobulin G4 (IgG4) monoclonal antibody that specifically binds to PD-1 molecules on the surface of T cells, thereby blocking the programmed death receptor-1 (PD-1)/programmed death receptor-1 ligand (PD-L1) pathway induced by tumor immune tolerance, and reactivating the antitumor activity of lymphocytes.

In summary, recurrence after radical treatment of liver cancer is an urgent clinical problem. Recurrent HCC treatment represented by resection, ablation and TACE is difficult to achieve more satisfactory efficacy. The main ablative techniques includes radiofrequency ablation, microwave ablation and cryoablation.As a local treatment for liver cancer, ablation has the risk of incomplete ablation and insufficient ablation margin, and because RFA cannot resolve micrometastases, tumor growth, invasion and metastasis occur. Therefore, ablation combined with lenvatinib and immune checkpoint inhibitors have theoretical complementary advantages, and this study intends to compare the clinical efficacy and safety of ablation combined with lenvatinib plus anti-PD-1 antibodies in the treatment of patients with early recurrent liver cancer compared with ablation alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, ≤75 years old, gender unlimited;
2. primary hepatocellular carcinoma proved pathologically and clinically;
3. 2 months after radical resection or ablation, imaging examination (MRI, CT plain enhanced) showed no tumor lesions, HCC recurred within 3 years after surgery, no extrahepatic metastasis;
4. ECOG score 0-1;
5. Recurrent liver cancer meets the Milan criteria: single tumor diameter ≤5cm or multiple tumors less than 3 with a maximum diameter ≤3cm, no major vascular invasion, no lymph node metastasis or extrahepatic metastasis;
6. Child-Pugh liver function grades: A, B;
7. Expected survival > 6 months;
8. Adequate organ function: ① no need for growth factors and blood components within 2 weeks prior to enrollment; (2) Cardiac function: no heart disease, coronary heart disease, cardiac function level 1-2; ③ In the first 7 days of enrollment, liver and kidney function was adequate and laboratory indicators were suitable (untreated) : HGB≧9.0g/dl, neutrophils ≧1,500/mm3, PLT≧50x109/L, serum ALB≧28g/L, TBIL<2mg /dL, ALT, AST< 5 times of the upper limit of normal value, Bun, Cr< 1.5 times of the upper limit of normal value, INR<1.7 or extended PT<3s;
9. Patients with normal blood pressure or hypertension should use antihypertensive drugs to control blood pressure within the normal range;
10. Diabetic patients should control fasting blood glucose ≤8mmol/L by hypoglycemic drugs;
11. No other serious diseases (such as autoimmune diseases, immune deficiency, organ transplantation, etc.) that conflict with the Plan;
12. No history of other malignant tumors;
13. Women of childbearing age must have a negative blood pregnancy test within seven days, and subjects of childbearing age must use appropriate contraception during the test and for six months after the test;
14. The patient agrees to participate in the clinical study and sign the Informed Consent.

Exclusion Criteria:

* (1) previous radiotherapy, hormone therapy or molecular targeted therapy; (2) Patients with distant metastasis confirmed by imaging; (3) The subject has had or co-has other malignancies (other than cured basal cell carcinoma of the skin and carcinoma in situ of the cervix); (4) The subject is known to be allergic to macromolecular protein preparations, or to any component of anti-PD-1 antibodies; (5) Subject has any history of active autoimmune disease or autoimmune disease (e.g., but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitaritis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; Subjects with childhood leukoplectic disease or complete remission of asthma can be incorporated into adults without any intervention; Subjects requiring medical intervention with bronchodilators are not included; (6) Subjects were taking immunosuppressants, or systemic or absorbable topical hormone therapy for immunosuppressive purposes (doses >10mg/ day of prednisone or other therapeutic hormones) and were still taking them within 2 weeks prior to enrollment; (7) Clinical symptoms of heart disease or disease not well controlled, such as: heart failure of grade 2 or above A.N. B. Unstable angina pectoris; C. Myocardial infarction within 1 year; D. Patients with clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention; (8) Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg>2g/L), bleeding tendency or receiving thrombolytic or anticoagulant therapy; (9) The patient has current (within 3 months) gastrointestinal conditions such as esophageal varices, active gastric and duodenal ulcers, ulcerative colitis, portal hypertension, or active bleeding from unexcised tumors, or other conditions identified by the investigator as likely to cause gastrointestinal bleeding and perforation; (10) Previous or current severe bleeding (bleeding >30 ml within 3 months), hemoptysis (fresh blood >5 ml within 4 weeks), or thromboembolic events (including stroke events and/or transient brain dysfunction) within 12 months; (11) Previous and current patients with objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-induced pneumonia, severe impairment of lung function, etc.; (12) of congenital or acquired immune deficiency, such as HIV infection, active hepatitis (transaminase does not meet the criteria for the hepatitis b reference: HBV DNA of 10 or higher ⁴ / ml; Hepatitis C reference: HCV RNA≥103/ml); Chronic hepatitis B virus carriers with HBV DNA<2000 IU/ml (<104 copies /ml) must also receive antiviral therapy during the trial to be enrolled; (13) Subjects are participating in other clinical studies or less than one month has passed since the end of the previous clinical study; Subjects may receive other systemic antitumor therapies during the study; (14) The subject is known to have a history of psychotropic, alcohol, or drug abuse; (15) Imaging examination confirmed tumor recurrence or metastasis 2 months after surgery; (16) The researcher believes that it should be excluded from this study. For example, in the researchers' judgment, the subjects had other factors that might have led to the study's termination, such as other serious medical conditions (including mental illness) requiring combination treatment. Serious laboratory abnormalities, accompanied by family or social factors, may affect the safety of the subject or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free Survival, RFS | 1 year
  Defined as the percentage of patients who had achieved 1 year of disease recurrence (i.e., intrahepatic recurrence or extrahepatic metastasis) or death (from any cause) from the date of enrollment, whichever occurred first.

SECONDARY OUTCOMES:
Recurrence free survival (RFS) at 2 years | 2 years
  Defined as the percentage of patients with no disease recurrence (i.e., intrahepatic recurrence or extrahepatic metastasis) or death (from any cause) for 2 years from the date of enrollment.
Recurrence free survival (RFS) at 3 years | 3 years
  Defined as the percentage of patients with no disease recurrence (i.e., intrahepatic recurrence or extrahepatic metastasis) or death (from any cause) for 3 years from the date of enrollment.
Safety: Incidence of adverse events | 18 months
  Incidence of adverse events, severe AES, death, and laboratory abnormalities in treated patients.
Overall Survival (OS) | 18 months
  Overall Survival (OS): defined as the time from randomization to death from any cause throughout the trial. Patients who drop out or are lost to follow-up will be treated as deleted, with the last known date of survival as the last time of survival. Patients still alive at the end of the study will also be treated as deleted, with the last known date of survival as the last survival time.
Recurrence free Survival (RFS) | 18 months
  Recurrence free Survival (RFS): defined as the time between recurrence of tumor or death (from any cause) after recurrence of HCC.
Biomarkers in tumors and peripheral blood | 18 months
  Biomarkers in tumor and peripheral blood such as AFP, CEA, CA199, CA125, RBC, Alb

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No